CLINICAL TRIAL: NCT04984044
Title: Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effect of Vitamin D in Patients With Diabetic Peripheral Neuropathy to Alleviate Pain and Improvement of Symptoms
Brief Title: Effect of Vitamin D in Patients With Diabetic Peripheral Neuropathy to Alleviate Pain and Improvement of Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Zannatul Ferdous, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2020/9630
Record Dates: First submitted 2021-05-30; First posted 2021-07-30 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: DPN; Vitamin D3; MNSI
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Diagnosed case of Type 2 Diabetes Mellitus with peripheral neuropathy
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): This arm includes 36 Diabetic Peripheral Neuropathy patients receiving the antidiabetic medications
  Interventions: Dietary Supplement: Vitamin D3
- Control (Placebo Comparator): This arm includes 36 Diabetic Peripheral Neuropathy patients receiving the antidiabetic medications
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Dietary supplement:Vitamin D3
  1 capsule of Vitamin D3 (40,000IU) weekly for 8 weeks with antidiabetic drug
  Other Names: Cholecalciferol
  Arms: Experimental
Dietary Supplement: Placebo — 1 capsule weekly for 8 weeks with antidiabetic drug
  Arms: Control

SUMMARY:
Diabetic peripheral neuropathy(DPN) is one of the major complications of diabetes mellitus which accelerates the occurrence of ulceration of diabetic foot and amputation of lower extremities as well as severely affects the quality of life. The treatment of this condition has remained unsatisfactory with a good response to conventional medications. It is now evident that vitamin D deficiency is common in diabetic patients and especially in these patients diagnosed with diabetic peripheral neuropathy. The present research is therefore designed to observe the effect of exogenous administration of vitamin D in diabetic peripheral neuropathy patients of Bangladesh.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy is one of the common complications of long-standing diabetes mellitus with a prevalence of 30% to 50%. It accelerates the occurrence of ulcers of diabetic foot and amputation of lower extremities as well as severely affects the quality of life. The treatment of this condition has remained unsatisfactory in spite of a good response to conventional medications. Studies showed that Vitamin D3 exerts a neuroprotective effect through the production of nerve growth factor (NGF) and neurotrophins. However, some recent trials demonstrated that vitamin D3 could be a promising agent in this regard. This proposed study was therefore an effort whether there is any role of vitamin D3 in improving symptoms of diabetic peripheral neuropathy patients. This study was a randomized, double-blind, placebo-controlled trial, conducted in the Department of Pharmacology in collaboration with the Department of Endocrinology of Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka from September 2019 to January 2022. A total of 72 patients suffering from diabetic peripheral neuropathy was enrolled according to inclusion and exclusion criteria. A validated version of the Michigan Neuropathy Screening Instrument (MNSI) and Visual Analogue Scale (VAS) was used to assess peripheral neuropathy. Then the patients were randomly allocated into two arms: control and intervention. The patient in the control arm received the standard antidiabetic medications plus one placebo capsule weekly orally for 8 weeks starting from the day of an initial assessment. On the other hand, the intervention arm received the standard antidiabetic medications plus one capsule of vitamin D3 (40,000 IU) weekly orally for 8 weeks starting from the day of an initial assessment. Data of HbA1c level was recorded and a blood sample was collected to measure serum 25(OH) D level at baseline and after 8 weeks of therapeutic intervention. Confirmation of the regular intake of medicine was ensured over the telephone, pill count, and from the patient's compliance sheet. After 8 weeks each patient was evaluated again using VAS and MNSI tools. Out of 72, 53 patients had completed the study and met the criteria for analysis. Therefore, Intention to Treat (ITT) was 72 and Per Protocol (PP) treatment was 53. The statistical tests used to analyze the data were the chi-square (x2) test, paired t-test, unpaired t-test, and Pearson correlation test. The chi-square (x2) test was used to compare categorical data between two groups. The independent t-test was used to compare the continuous data between two groups. P-value ≤ 0.05 was considered significant. After 8 weeks of treatment, the VAS score of pain in DPN patients in the intervention arm reduced significantly (P=0.00) from 5.50 ± 0.64 to 4.23 ± 0.98. In the intervention arm, statistically significant improvement was also observed in the MNSI score both for the questionnaire (from 8.54 ± 1.15 to 6.00 ± 1.32; P=0.00) and physical assessment (from 3.44 ± 1.22 to 2.40 ± 1.06; P=0.00) respectively. Serum 25(OH)D level significantly improved (P=0.00) after oral administration of vitamin D3 in the intervention arm from 10.83 ± 4.47 ng/ml to 17.79 ± 7.53 ng/ml. The reduction observed in HbA1c level in the intervention arm (from 8.66 ± 1.39 to 7.25 ± 0.87) was significant (P=0.00). This should be noted that a significant reduction of VAS score (P= 0.04) and MNSI questionnaire score (P=0.00) was observed in the placebo arm after 8 weeks, though the difference between the reduction achieved was significant between placebo and intervention arm (for VAS, P=0.00 and for MNSI, P=0.00). However, in the control arm, there was no significant reduction (P=0.69) in MNSI physical assessment score. A negative correlation was observed between serum 25(OH) D level and VAS (r= -0.1) and MNSI score (r= -0.17) respectively. Oral administration of 40,000 IU vitamin D3 weekly for 8 weeks along with standard antidiabetic medications produces a significant reduction of the level of pain and other neuropathic symptoms in the patients with Diabetic Peripheral Neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type II Diabetes Mellitus patients who have been on anti-diabetic therapy for 1 year or more
* Diabetic patient who meet the clinical criteria for DPN diagnosed by an endocrinologist of OPD of endocrinology
* Age between 30 and 70 years
* Gender: Both Male and Female
* Patients who will give informed written consent

Exclusion Criteria:

* Patients suffering from other causes of peripheral neuropathy for example chemotherapy-induced neuropathy, hyperthyroidism or hypothyroidism, rheumatoid arthritis, SLE
* Pregnant or lactating women
* Patients with renal and liver disease, psychiatric disorder
* Patients receiving vitamin D, vitamin B6, vitamin B12 supplementation, anticonvulsants, antidepressants, opioids, and other neuropathic pain medications within the last two months.
* Serum calcium level: > 10.2 mg/dl
* HbA1c level > 11%

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Visual Analogue Scale(VAS) score at 8 weeks. | 8 weeks
  Assessment of severity of pain by using Visual Analogue Scale(VAS) at baseline and after 8 weeks and compare the score between two groups. VAS is a 0-10 numeric pain scale scored by No pain (score 0-3), moderate pain (scoring 4-6), and unbearable pain (score 7-10).
Change from baseline Michigan Neuropathy Screening Instrument (MNSI) scores at 8 weeks. | 8 weeks
  Assessment of severity of neuropathic symptoms by using MNSI score at baseline and after 8 weeks and comparing the score between two groups. MNSI is composed of 15 items questionnaire and a brief clinical examination. MNSI questionnaire score of 7 or more indicates the presence of diabetic peripheral neuropathy. 13 is the highest score indicating the worst disease. Whereas, MNSI Physical assessment score of 2.5 or more indicates the presence of diabetic peripheral neuropathy.

SECONDARY OUTCOMES:
Change from baseline Serum 25(OH) D level at 8 weeks. | 8 weeks
  Serum 25(OH) D level is assessed at baseline and 8 weeks following vitamin D administration. Compare the serum 25(OH) D level between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zannatul Ferdous, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Prof. Md. Sayedur Rahman, MBBS, M Phil, FCPS, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Department of Pharmacology, BSMMU, Dhaka, Bangladesh